CLINICAL TRIAL: NCT00840125
Title: A Phase II Open-Label Study Designed to Evaluate the Efficacy and Safety, of Erlotinib in Combination With Docetaxel in Selected Non Small Cell Lung Cancer Patients Eligible for First Line Treatment
Brief Title: Study of Erlotinib With Docetaxel in Selected Non Small Cell Lung Cancer Patients in First Line Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG-NSCLC-2008
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; ERLOTINIB; DOCETAXEL; first line treatment; Stage IIIB /IV; not previously treated; ECOG PS 2 or age over 65
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): docetaxel + erlotinib
  Interventions: Drug: erlotinib; Drug: docetaxel

INTERVENTIONS:
Drug: erlotinib — 150mg tablet daily
  Other Names: tarceva
Drug: docetaxel — 30 mg/m2 days 1,8 of 22 days cycles, up to 6 cycles
  Other Names: taxotere

SUMMARY:
Study Rationale:

There is increasing evidence that erlotinib improves overall survival in selected patients with stage IIIB-IV NSCLC. Furthermore, pre-clinical and phase II studies have shown a potential for synergism between erlotinib and docetaxel. This study will further evaluate the effects of combination treatment on overall survival in selected NSCLC patient population.

Based on recent published data, the treatment cycle in this study will be 22 days with two infusions (Day 1 and Day 8 of each cycle). This is different from the standard therapy care of 28-day cycle (three infusions on Days 1, 8 and 15). The shorter 22-day cycle was shown to be just as effective as the 28-day cycle and is expected to increase subject compliance and decrease chemotherapy-induced toxicity.

Study Objectives:

The primary objective is to demonstrate superiority in progression-free-survival, when erlotinib is added to docetaxel.

The secondary objectives are to determine:

* Overall survival (defined as the time period from the start of first-line therapy to death)
* Time to treatment failure or disease progression (defined as the time period from the start of first-line therapy to investigator assessed disease progression)
* Tumor response rate and duration
* Safety profile
* Quality of Life improvement
* microRNA profile (assessed from human lung biopsy and/or cytology samples) at screening for prognostic purposes

DETAILED DESCRIPTION:
Study Design:

This will be a Phase II, open-label, single-center, repeat dose, study. After a two-week screening phase, eligible subjects will receive combined docetaxel and erlotinib treatment over six cycles. Each 22-day treatment cycle will consist of two infusion of docetaxel, one-week apart followed by one week rest, and daily administration of erlotinib. Subjects, who complete six cycles of combination therapy, will continue receiving erlotinib monotherapy for as long as they are benefiting from this therapy in the opinion of the investigator (i.e. until continued toxicity or disease progression or withdrawal from the study). Subjects will be evaluated for safety and radiologic tumor assessment throughout the study until death. The study will be terminated after every living patient has had a follow up of at least 6 months after stopping TarcevaTM, or when all patients have died.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, above 18 years of age at the time of enrollment.
2. Subject aged 18-65 must have ECOG performance status of 2 and subjects above 65 must have ECOG PS 0-2.
3. Histological or cytological documented diagnosis of inoperable, locally advanced (with pleural effusion), recurrent or metastatic (Stage IIIB or Stage IV) NSCLC.
4. Patients must have evidence of measurable disease with at least one measurable or evaluable lesion.
5. Eligible for first line monotherapy treatment (or no prior chemotherapy or radiation treatments for this indication). Palliative localized radiation is allowed.
6. Life expectancy of at least 12 weeks.
7. Adequate bone marrow function as shown by: WBC >= 3.0 x 109/L, ANC >=1.5 x 109/L, Platelets >=100 x 109/L, Hgb >=10g/dL.
8. Subjects must have normal organ function as defined below:

   * AST (SGOT) / ALT (SGPT) ≤ 2 x upper limit of normal (ULN),
   * Serum creatinine ≤ 1.5 x ULN or creatinine clearance > 60 ml/min
   * Coagulation markers - PT and PTT (or INR) within normal limits unless subjects are already anti-coagulated for other reasons (i.e., atrial fibrillation, etc.).
9. Signed written informed consent to participate in the study.
10. Ability to comply with the requirements of the study.

Exclusion Criteria:

1. Participation in an investigational trial within 30 days of the screening visit.
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib or docetaxel.
3. Have a previous (unless disease free for more than five years) or concurrent malignancy besides NSCLC (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer).
4. Subjects with known brain metastases or spinal cord compression that is newly diagnosed and/or has not yet been definitively treated with surgery and/or radiation; previously diagnosed and treated CNS metastases or spinal cord compression with evidence of stable disease (clinically stable imaging) for at least 2 months is permitted..
5. Subjects with preexisting neuropathy ≥ grade 2.
6. Current serious infections.
7. Current known acute or chronic infection with HBV or HCV.
8. Known human immunodeficiency virus (HIV) infection.
9. Any significant ophthalmologic abnormality, especially severe dry eye syndrome, keratoconjunctivitis sicca, Sjögren syndrome, severe exposure keratitis or any other disorder likely to increase the risk of corneal epithelial lesions. The use of contact lenses is not recommended during the study. The decision to continue to wear contact lenses should be discussed with the patient's treating Oncologist and the ophthalmologist.
10. Subjects with other concurrent severe and/or uncontrolled medical condition which could compromise participation in the study (i.e. active infection, uncontrolled diabetes, uncontrolled hypertension - grade 4, congestive cardiac failure, unstable angina, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, chronic liver or renal or metabolic disease, active upper GI tract ulceration).
11. Any chronic or acute condition susceptible of interfering with the evaluation of drug effect.
12. Any form of substance abuse (including drug or alcohol abuse), psychiatric disorder or any chronic condition susceptible, in the opinion of the investigator, of interfering with the conduct of the study.
13. Organ allograft or previous history of stem cell transplantation.
14. Subjects who received anti-neoplastic therapy, radiation therapy or had surgery within 28 days prior to the start of study agent administration or who have not recovered from the toxic effects of such therapy. Palliative localized radiation is allowed.
15. Subjects who cannot take oral medication, who require intravenous alimentation, have had prior surgical procedures affecting absorption, or have active peptic ulcer disease.
16. Fertile subjects who are not willing to use an acceptable method of contraception during the treatment period and for 28 days following completion of treatment.
17. For women of child-bearing potential: A positive pregnancy test at screening or breast-feeding.
18. Subjects who are likely to be non-compliant or uncooperative during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Maya Gottfried, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel, Israel